"Evaluation of The Effect of Neck and Trunk Stabilization Exercises on Quality of Life and Communication in Children with Cerebral Palsy with Oral Motor Problem"

NCT04214080

03.12.2019

## **Statistical Analysis Plan**

Descriptive statistics for continuous variables are expressed as mean (X), standard deviation (SD) values (Height, weight, body mass index (BMI), gender, etc); it is expressed as number (n) and percentage (%) for categorical variables.

In calculations, statistical significance level ( $\alpha$ ) was taken as 5% and values with p<0.05 expressed statistical significance. "Statistical Package for Social Sciences" (SPSS 16) statistics program was used for calculations.

Non-parametric tests were applied since the continuous variables in the study were not normally distributed. Mann-Whitney U test was used to compare continuous variables according to Control and Study groups (Visual Analogue Scale, Viking Speech Scale, Communication Function Classification System, Katz scale, Sub-parameters of PedsQL). Wilcoxan test was used for intra groups comparisons (Visual Analogue Scale, Viking Speech Scale, Katz scale, Sub-parameters of PedsQL). In determining the relationship between categorical variables and groups, Chi-square test was performed (CP subtypes, Number of Medication, Types of Medications).

Spearman's Correlation Analysis was used to determine the relationship between groups of cases and other categorical and continuous variables (Visual Analogue Scale and Katz scale correlation analysis results with Communication Function Classification Systems).